CLINICAL TRIAL: NCT04375722
Title: Exogenous Tuning of Neural Oscillations as a Mode of Treatment in Post-stroke Aphasia
Brief Title: Transcranial Alternating Current Stimulation (tACS) in Aphasia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Priyanka Shah-Basak, PhD, Priyanka Shah-Basak, PhD, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 36878
Record Dates: First submitted 2020-05-01; First posted 2020-05-05 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Aphasia; Stroke
Keywords: language; language impairment; transcranial alternating current stimulation; tACS
MeSH Terms: conditions — Aphasia; Stroke; Language; Language Disorders

STUDY DESIGN:
Intervention Model Description: In the within-subject design healthy participants and stroke survivors will receive tACS stimulation with active and/or sham settings in a randomized order with >48 hours washout period in between stimulation sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- tACS 10 Hz low frequency (Experimental): All participants in a within-subject design will receive high-Definition-tACS, delivered via a battery operated alternating current stimulator (Soterix) using two 3x1 center-surround montages. Targets of stimulation will be localized based on the 10-10 International EEG system with center electrodes placed at a frontal and a temporoparietal site. The current is turned on and increased in a ramplike fashion over approximately 30 seconds. Participants will undergo tACS with frequencies ranging from 4-40Hz for 20-minutes with 2 milliampere (mA) peak-to-peak intensity. For sham stimulation, tACS is turned off after the first 30 seconds.
  Interventions: Device: tACS

INTERVENTIONS:
Device: tACS — Active or Sham tACS will be applied.

SUMMARY:
This study will assess the effects of transcranial alternating current stimulation (tACS) on language recovery after stroke as well as healthy language functions.

DETAILED DESCRIPTION:
Aphasia is a debilitating disorder, typically resulting from damage to the left hemisphere, that can impair a range of communication abilities, including language production and comprehension, reading, and writing. Approximately 180,000 new cases of aphasia are identified per year, and approximately 1 million or 1 in 250 are living with aphasia in the United States (NIH-NIDCD, 2015). Treatments are limited and provide modest benefits at best. The current emphasis in aphasia rehabilitation is to formulate intensive speech and language therapies and augment therapeutic benefits by providing brain stimulation concurrent with therapies.

The current study will investigate the efficacy of high-definition tACS (HD-tACS) to help restore neural oscillatory activity in aphasia. TACS differs from widely used transcranial direct current stimulation (tDCS) in that sinusoidal, alternating currents are delivered rather than constant currents. TACS can manipulate the ongoing oscillatory neuronal activity and potentially increase functional synchronization (or connectivity) between targeted areas. This feature of tACS is quite attractive, given the new body of evidence suggesting that language impairments stem from diminished functional connectivity and disruptions in the language network due to stroke. The selection of tACS frequencies in this study is guided by our preliminary work examining pathological neural oscillations found near stroke-lesioned areas (or perilesional) in aphasia and by the involvement of specific frequencies during a verbal short-term memory task. By exogenously tuning the neural oscillations with tACS, the investigators hope to up-regulate communication across regions within the language network and other connected areas to improve outcomes. If successful, tACS will be a powerful and novel treatment approach with reverberating positive impact on long-term recovery.

The study will employ HD-tACS in a within-subject and sham-controlled design, using frequencies ranging from theta to low-gamma (4-40 Hz) combined with language tasks. Magnetoencephalography (MEG) or electroencephalography (EEG) will be used to determine tACS frequencies and to evaluate behavioral and neurophysiological changes in response to tACS. Investigators plan to recruit 200 participants: 100 stroke survivors with aphasia and 100 healthy controls.

Participants will complete language testing that covers a broad range of language functions, medical history, and MRI. Eligible participants will undergo active tACS or sham-tACS over 3-4 sessions. The tACS administrator and participants will be blinded to the stimulation type. The order of stimulation type will be counterbalanced across participants. Washout period between visits will be at least 48 hours to minimize potential carryover effects. MEG will be collected prior to tACS sessions during a language task to determine tACS frequency. EEG may be acquired before and after tACS during periods of rest (resting-state) and during language tasks. Participants will complete a questionnaire at the end of stimulation visits to assess potential side effects of tACS. Total time enrolled in the study is expected to be 2-3 weeks, which may be longer depending on participant's availability.

ELIGIBILITY:
Inclusion Criteria:

Healthy Controls

* 18 years of age or older
* Fluent in English
* No history of neurological or psychiatric disorders

Stroke Patients

* Diagnosed with post-stroke aphasia by referring physician/neuropsychologist
* Consent date >=1 months after stroke onset
* Right-handed
* Fluent in English
* 18 years of age or older

Exclusion Criteria:

* Severe cognitive, auditory or visual impairments that would preclude cognitive and language testing
* Presence of major untreated or unstable psychiatric disease
* A chronic medical condition that is not treated or is unstable
* The presence of cardiac stimulators or pacemakers
* Any metal implants in the skull
* Contraindications to MRI or tACS
* History of seizures
* History of dyslexia or other developmental learning disabilities

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-01-04 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
tACS changes in language performance verbal STM tasks | Changes monitored over pre, during and immediately after 20 minutes of tACS
  Improvement on verbal STM performance as determined by increases in span, accuracy or decreases in reaction time is expected with active tACS.
tACS-dependent neurophysiological changes | Changes monitored over pre and immediately after 20 minutes of tACS
  Concomitant frequency-specific EEG changes in spectral power and phase synchronization are expected.

SECONDARY OUTCOMES:
Individual differences in tACS responsiveness | Based on immediate changes monitored after 20 minutes of tACS
  tACS responsiveness depending on language impairment types, stroke lesion and language lateralization characteristics will be explored.

CONTACTS AND LOCATIONS:
Overall Officials: Priyanka Shah-Basak, PhD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antal A, Alekseichuk I, Bikson M, Brockmoller J, Brunoni AR, Chen R, Cohen LG, Dowthwaite G, Ellrich J, Floel A, Fregni F, George MS, Hamilton R, Haueisen J, Herrmann CS, Hummel FC, Lefaucheur JP, Liebetanz D, Loo CK, McCaig CD, Miniussi C, Miranda PC, Moliadze V, Nitsche MA, Nowak R, Padberg F, Pascual-Leone A, Poppendieck W, Priori A, Rossi S, Rossini PM, Rothwell J, Rueger MA, Ruffini G, Schellhorn K, Siebner HR, Ugawa Y, Wexler A, Ziemann U, Hallett M, Paulus W. Low intensity transcranial electric stimulation: Safety, ethical, legal regulatory and application guidelines. Clin Neurophysiol. 2017 Sep;128(9):1774-1809. doi: 10.1016/j.clinph.2017.06.001. Epub 2017 Jun 19. PMID 28709880
- [Background] Bucur M, Papagno C. Are transcranial brain stimulation effects long-lasting in post-stroke aphasia? A comparative systematic review and meta-analysis on naming performance. Neurosci Biobehav Rev. 2019 Jul;102:264-289. doi: 10.1016/j.neubiorev.2019.04.019. Epub 2019 May 8. PMID 31077693
- [Background] Buzsaki, G. (2006). Rhythms of the brain. New York: Oxford.
- [Background] Chu RK, Braun AR, Meltzer JA. MEG-based detection and localization of perilesional dysfunction in chronic stroke. Neuroimage Clin. 2015 Apr 8;8:157-69. doi: 10.1016/j.nicl.2015.03.019. eCollection 2015. PMID 26106540
- [Background] Dubovik S, Ptak R, Aboulafia T, Magnin C, Gillabert N, Allet L, Pignat JM, Schnider A, Guggisberg AG. EEG alpha band synchrony predicts cognitive and motor performance in patients with ischemic stroke. Behav Neurol. 2013;26(3):187-9. doi: 10.3233/BEN-2012-129007. PMID 22713421
- [Background] Finnigan S, van Putten MJ. EEG in ischaemic stroke: quantitative EEG can uniquely inform (sub-)acute prognoses and clinical management. Clin Neurophysiol. 2013 Jan;124(1):10-9. doi: 10.1016/j.clinph.2012.07.003. Epub 2012 Aug 2. PMID 22858178
- [Background] Finnigan SP, Walsh M, Rose SE, Chalk JB. Quantitative EEG indices of sub-acute ischaemic stroke correlate with clinical outcomes. Clin Neurophysiol. 2007 Nov;118(11):2525-32. doi: 10.1016/j.clinph.2007.07.021. Epub 2007 Sep 21. PMID 17889600
- [Background] Fridriksson J, Rorden C, Elm J, Sen S, George MS, Bonilha L. Transcranial Direct Current Stimulation vs Sham Stimulation to Treat Aphasia After Stroke: A Randomized Clinical Trial. JAMA Neurol. 2018 Dec 1;75(12):1470-1476. doi: 10.1001/jamaneurol.2018.2287. PMID 30128538
- [Background] Fries P. Rhythms for Cognition: Communication through Coherence. Neuron. 2015 Oct 7;88(1):220-35. doi: 10.1016/j.neuron.2015.09.034. PMID 26447583
- [Background] Grefkes C, Fink GR. Reorganization of cerebral networks after stroke: new insights from neuroimaging with connectivity approaches. Brain. 2011 May;134(Pt 5):1264-76. doi: 10.1093/brain/awr033. Epub 2011 Mar 16. PMID 21414995
- [Background] Helfrich RF, Schneider TR, Rach S, Trautmann-Lengsfeld SA, Engel AK, Herrmann CS. Entrainment of brain oscillations by transcranial alternating current stimulation. Curr Biol. 2014 Feb 3;24(3):333-9. doi: 10.1016/j.cub.2013.12.041. Epub 2014 Jan 23. PMID 24461998
- [Background] Herrmann CS, Rach S, Neuling T, Struber D. Transcranial alternating current stimulation: a review of the underlying mechanisms and modulation of cognitive processes. Front Hum Neurosci. 2013 Jun 14;7:279. doi: 10.3389/fnhum.2013.00279. eCollection 2013. PMID 23785325
- [Background] Kielar A, Deschamps T, Chu RK, Jokel R, Khatamian YB, Chen JJ, Meltzer JA. Identifying Dysfunctional Cortex: Dissociable Effects of Stroke and Aging on Resting State Dynamics in MEG and fMRI. Front Aging Neurosci. 2016 Mar 3;8:40. doi: 10.3389/fnagi.2016.00040. eCollection 2016. PMID 26973515
- [Background] Shah-Basak PP, Wurzman R, Purcell JB, Gervits F, Hamilton R. Fields or flows? A comparative metaanalysis of transcranial magnetic and direct current stimulation to treat post-stroke aphasia. Restor Neurol Neurosci. 2016 May 2;34(4):537-58. doi: 10.3233/RNN-150616. PMID 27163249
- [Background] Shah-Basak PP, Kielar A, Deschamps T, Verhoeff NP, Jokel R, Meltzer J. Spontaneous oscillatory markers of cognitive status in two forms of dementia. Hum Brain Mapp. 2019 Apr 1;40(5):1594-1607. doi: 10.1002/hbm.24470. Epub 2018 Nov 12. PMID 30421472
- [Background] Shah-Basak PP, Norise C, Garcia G, Torres J, Faseyitan O, Hamilton RH. Individualized treatment with transcranial direct current stimulation in patients with chronic non-fluent aphasia due to stroke. Front Hum Neurosci. 2015 Apr 21;9:201. doi: 10.3389/fnhum.2015.00201. eCollection 2015. PMID 25954178